CLINICAL TRIAL: NCT01911156
Title: Sustained Off-treatment Response After HBeAg Loss in HBeAg-Pos Chronic Hepatitis B Patients Treated With Nucleos(t)Ide Analogues
Brief Title: Sustained Off-treatment Response After HBeAg Loss in Chronic Hepatitis B Patients Treated With Nucleos(t)Ide Analogues
Acronym: Stop
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stop Study; GILEAD Sciences Canada, Inc. (Other Grant/Funding Number: GILEAD Sciences Canada, Inc.)
Record Dates: First submitted 2013-06-25; First posted 2013-07-30 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Discontinue NA treatment (Other): Subjects will not receive NA during the 72 week study period
  Interventions: Drug: Discontinue NA Treatment
- NA treatment (Other): Subjects will continue to receive their prescribed NA during the 72 week study period
  Interventions: Drug: Continue NA treatment

INTERVENTIONS:
Drug: Continue NA treatment — Prescribed NA during the 72 week study period
  Arms: NA treatment
Drug: Discontinue NA Treatment — Discontinue NA Treatment
  Arms: Discontinue NA treatment

SUMMARY:
This is a prospective randomized, open-label, phase IV clinical trial to learn the effects, good and/or bad, of discontinuing or continuing nucleos(t)ide analogue (NA) treatment for 72 weeks in participants with chronic hepatitis B infection whose immune system is controlling the amount of virus levels in the blood for at least 12 months of NA therapy.

About 66 adult men and women will participate in this study from University Health Network which includes the Toronto Western Hospital for about 72 weeks.

DETAILED DESCRIPTION:
Chronic infection with the hepatitis B virus (HBV) is prevalent world-wide (estimated to affect 360 million individuals).

Chronic hepatitis b may result in progressive liver disease that leads to cirrhosis, end-stage liver disease and hepatocellular carcinoma (HCC). Chronic hepatitis B can also be benign and non-progressive, evolving into an inactive carrier state that rarely leads to significant liver injury or HCC. Over the last few years, several highly effective antiviral agents have been developed and approved for use in the treatment of chronic hepatitis B. Current therapy of chronic hepatitis B (CHB) aims at stopping progression to cirrhosis and hepatocellular carcinoma.

This is a prospective randomized, open-label, phase IV clinical trial to learn the effects, good and/or bad, of discontinuing or continuing NA treatment for 72 weeks in participants with chronic hepatitis B infection whose immune system is controlling the amount of virus levels in the blood for at least 12 months of NA therapy.

About 66 adult men and women will participate in this study from University Health Network which includes the Toronto Western Hospital for about 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B (HBsAg positive > 6 months)
* Currently on NA monotherapy and for ≥1 year prior to screening
* HBeAg negative with anti-HBe antibodies and HBV DNA undetectable at least once at 12 or more months prior to screening and at screening (HBV DNA assay should have lower limit of quantification of at least 50 IU/mL)
* Documented HBeAg positive before start of NA monotherapy
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Treatment with any investigational drug within 30 days of screening
* Severe hepatitis activity as documented by ALT >10x ULN
* Creatinine clearance <70 ml/min
* Presence of cirrhosis as documented by biopsy within 5 years, fibroscan >9kPa, or fibrotest >0.48
* Pre-existent neutropenia (neutrophils ≤1,000/mm3)
* Co-infection with hepatitis C virus and/or human immunodeficiency virus (HIV)
* Other acquired or inherited causes of liver disease
* Alpha fetoprotein >50 ng/ml
* Hyper- or hypothyroidism
* Immune suppressive treatment within the previous 6 months
* Pregnancy, lactation
* Other significant medical illnesses that might interfere with this study
* Any medical condition requiring, or likely to require chronic systemic administration of steroids, during the course of the study
* Substance abuse (alcohol (≥80 g/day)and inhaled drugs (past 2 years)
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Sustained response, defined as the presence of an HBV DNA level <2000 IU/ml at week 48 in patients with a combined response at baseline | Outcome of patients in whom NA monotherapy is stopped at week 0 and of patients who continue to receive NA monotherapy up till week 72

CONTACTS AND LOCATIONS:
Overall Officials: Harry Janssen, Prof., Principal Investigator — University Heath Network
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Dongelmans EJ, Feld JJ, Boonstra A, Brakenhoff SM, Wong D, Yim C, Claassen M, Honkoop P, Hansen BE, de Man RA, Fung S, Berg T, van Bommel F, Janssen HLA, Sonneveld MJ. Early HBcrAg and Anti-HBc Levels Identify Patients at High Risk for Severe Flares After Nucleos(t)ide Analogue Cessation-A Pooled Analysis of Two Clinical Trials. Aliment Pharmacol Ther. 2025 Feb;61(3):570-578. doi: 10.1111/apt.18416. Epub 2024 Dec 3. PMID 39624922
- [Derived] Liem KS, Chi H, Fung S, Wong DK, Yim C, Noureldin S, Chen J, de Man RA, Sarowar A, Feld JJ, Hansen BE, Hou J, Peng J, Janssen HLA. Early virologic relapse predicts alanine aminotransferase flares after nucleos(t)ide analogue withdrawal in patients with chronic hepatitis B. J Viral Hepat. 2022 Nov;29(11):986-993. doi: 10.1111/jvh.13742. Epub 2022 Sep 14. PMID 36048970
- [Derived] Liem KS, Fung S, Wong DK, Yim C, Noureldin S, Chen J, Feld JJ, Hansen BE, Janssen HLA. Limited sustained response after stopping nucleos(t)ide analogues in patients with chronic hepatitis B: results from a randomised controlled trial (Toronto STOP study). Gut. 2019 Dec;68(12):2206-2213. doi: 10.1136/gutjnl-2019-318981. Epub 2019 Aug 28. PMID 31462554